CLINICAL TRIAL: NCT05342064
Title: Closing -TB GAPs - for People Living With HIV: TB Guidance for Adaptable Patient-Centered Service
Acronym: TB_GAPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); London School of Hygiene and Tropical Medicine (Other); University of Ottawa (Other); University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Anna Mandalakas, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: H-51421
Record Dates: First submitted 2022-03-03; First posted 2022-04-22 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Tuberculosis; HIV Coinfection; Tuberculosis Infection
Keywords: TB/HIV co-infection; pediatric tuberculosis; tuberculosis preventive therapy
MeSH Terms: conditions — Tuberculosis; HIV Infections; Latent Tuberculosis

STUDY DESIGN:
Intervention Model Description: The study will be implemented within a non-randomized stepped-wedge pragmatic intervention study design with nested randomized screening, diagnostic and adherence studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (No Intervention): No intervention will be administered. Observational data regarding TPT uptake and adherence will be captured on all participants presenting for care
- TB screening and evaluation followed by TPT via a decentralized delivery system (Experimental): The intervention phase includes i) enrolling participants who have had TB disease excluded and allowing participant selection of a preferred TPT regimen, and ii) randomizing participants to one of two participant adherence support modalities.
  Interventions: Other: patient-centered TB preventive therapy; Other: TB preventive therapy adherence support

INTERVENTIONS:
Other: patient-centered TB preventive therapy — The intervention phase includes i) enrolling participants who have had TB disease excluded and allowing participant selection of a preferred TPT regimen, and ii) randomizing participants to one of two participant adherence support modalities.
  Arms: TB screening and evaluation followed by TPT via a decentralized delivery system
Other: TB preventive therapy adherence support — As part of this study, enhanced adherence support will be provided via bi-directional messaging and/or via clinic phone calls. All participants randomized to enhanced adherence support will receive a weekly text reminder beginning seven days after the initiation. Each message will ask participants if they would like to be contacted to discuss any questions and will prompt participants to ask questions by text if more convenient or preferable. All text-based questions from participants will be answered by a trained nurse with back up from a physician.
  Arms: TB screening and evaluation followed by TPT via a decentralized delivery system

SUMMARY:
Tuberculosis (TB) is the world's leading infectious cause of mortality and responsible for 1/3 of deaths in people living with human immunodeficiency virus (PLHIV). Children and adolescents living with HIV (CALHIV) are disproportionately affected due to inadequate preventive services, large case detection gaps, treatment and adherence challenges, and knowledge gaps. This project will generate evidence to inform interventions targeting several of these weaknesses in the TB/HIV cascade of care.

Early detection and treatment of TB improve outcomes in people living with HIV (PLHIV). A key challenge in the detection of HIV-associated TB has been the implementation of screening that identifies the correct population for diagnostic testing. Increasing evidence demonstrates the poor performance of recommended symptom screens and diagnostic approaches. Hence, the investigators aim to define a more accurate TB screening and testing strategy among PLHIV (Objective 1 and Objective 2).

TB preventive treatment (TPT) averts HIV-associated TB. Nevertheless, among PLHIV, TPT initiation and completion rates are sub-optimal and effective delivery strategies are not defined. As such, the investigators aim to identify the most effective TPT delivery strategy through shared decision making and by integrating approaches proven to be effective at improving HIV treatment adherence (Objective 3).

Although evidence demonstrates that isoniazid preventive therapy (IPT) is cost-effective in young children living in TB/HIV high burden settings, the cost-effectiveness of newer short-course TPT has primarily been studied in the context of a TB low-burden, high-income setting. The investigators aim to generate evidence to fill this knowledge gap and inform policy for PLHIV living in TB/HIV high burden settings (Objective 4).

This study is supported by the Centers for Disease Control and Prevention of the U.S. Department of Health and Human Services (HHS) as part of a financial assistance award totaling an anticipated $5,000,000 over five years with 100 percent funded by CDC/HHS.

ELIGIBILITY:
OBJECTIVES 1 and 2:

Inclusion Criteria:

* HIV positive or HIV exposed and presumptively positive while awaiting confirmatory testing in infants

Exclusion Criteria:

* do not provide informed consent or assent as appropriate or are currently being treated for TB

OBJECTIVE 3:

Inclusion Criteria:

* negative TB symptom screen OR for whom TB disease has been ruled out in accordance with WHO Guidelines in adults and according to consensus definitions for child TB

Exclusion Criteria:

* do not provide informed consent or assent as appropriate or are currently being treated for TB

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6500 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
TB screening | 24-32 months
  Sensitivity of C-reactive protein for TB screening compared to the sensitivity of the WHO symptom screening using the McNemar test
TB diagnosis | 24-32 months
  Sensitivity of Xpert Host Response Cartridge compared with the sensitivity of Xpert Ultra on sputum or on gastric aspirate using the McNemar test
TPT prevention outcomes | 48 months
  Comparing TPT completion rates in participants randomized to bi-directional messaging support vs. standard support
Cost-effectiveness | 32 months
  Estimating the incremental cost-effectiveness of new shortened TPT regimens measured as cost per DALYS averted for each TPT strategy and the enhanced participant support modality compared with current standard of care

SECONDARY OUTCOMES:
Proportion of participants selecting 3HP and the proportion selecting 6H when offered a choice within a decentralized model | 48 months
Proportion of participants completing 6H and the proportion completing 3HP among participants randomized to standard support vs. bidirectional messaging | 48 months
  Treatment completion will be defined as receipt of at least 80% of doses during a pre-specified period of time and consistent with WHO definitions.
Proportion of participants initiated on TPT in the control phase vs. the intervention phase | 48 months
  Initiation rates will be estimated by the number of participants initiating TPT divided by the number of instances that TPT was offered
Description of the number of participants with different TB treatment and TPT outcomes at the completion of respective therapies | 48 months
  At individual study end point or at study closure, participants will be classified as i) retained in care, ii) died, iii) lost to follow-up, or iv) transferred out.
Number of life years saved through novel TPT approaches | 32 months
Number of active TB cases averted through novel TPT approaches | 32 months
Measure the association between participant factors and screening and diagnostic positivity rates | 24-32 months
  Participant factors are inclusive but not limited to TB infection status, immunologic, virologic, demographic, socioeconomic and clinical factors. The screening and diagnosis approaches are: point of care C-reactive protein, chest radiography, Fuji-LAM, Xpert Ultra performed on oral swabs and stool specimens and ultrasound.
Laboratory turnaround time | 24-32 months
  For all screening and diagnostic tests of the study
Result reporting rate | 24-32 months
  For all screening and diagnostic tests of the study
Time-to-treatment initiation | 24-32 months
  For all screening and diagnostic tests of the study
Diagnostic performance of mask sampling with differing forms of quiet and forced expiration (i.e., talking, singing) against standard approaches of sampling | 24-32 months
Compare alternative stool processing techniques and molecular diagnostics/tests of MTB resistance against clinical and microbiologic reference standards | 24-32 months
  Done using de-identified stool collected and bio-banked during the study.
Compare Alere-LAM diagnostic accuracy with that of the SILVAMP-LAM with both spot and early-morning urine samples | 24-32 months
Analyze different processing approaches for oral swabs prior to testing by Xpert Ultra vs. other microbiological diagnostic and drug susceptibility tests | 24-32 months
Compare clinician read of chest radiograph with point-of-care ultrasound interpretation to determine agreement and additive yield of each method | 24-32 months
  this outcome will be studied only in Eswatini and Malawi
Prevalence of extrapulmonary TB by means of point of care ultrasound in participants diagnosed with TB | 24-32 months
Assess ultrasound inter-reader agreement between hands-on operators | 24-32 months
Assess ultrasound inter-reader agreement between hands-on operators AND remote expert reviewers | 24-32 months
Compare the proportion of clinician and computer aided detection chest radiograph interpretation with algorithmic approaches against clinical and microbiologic reference standards | 24-32 months
Sensitivity of point of care CRP versus the WHO symptom screening | 24-32 months
  CRP will be performed on whole blood using the FDA approved POC iChroma assay. A CRP of > 10 mg/L will be considered positive
Specificity of point of care CRP versus the WHO symptom screening | 24-32 months
  CRP will be performed on whole blood using the FDA approved POC iChroma assay. A CRP of > 10 mg/L will be considered positive
Area under the receiver operator curve of point of care CRP versus the WHO symptom screening | 24-32 months
  CRP will be performed on whole blood using the FDA approved POC iChroma assay. A CRP of > 10 mg/L will be considered positive
Sensitivity of chest radiography versus the WHO symptom screening | 24-32 months
  Chest radiography will be interpreted as normal or abnormal for the purposes of TB screening and will be evaluated using a standardized interpretation form
Area under the receiver operator curve of chest radiography versus the WHO symptom screening | 24-32 months
  Chest radiography will be interpreted as normal or abnormal for the purposes of TB screening and will be evaluated using a standardized interpretation form
Specificity of chest radiography versus the WHO symptom screening | 24-32 months
  Chest radiography will be interpreted as normal or abnormal for the purposes of TB screening and will be evaluated using a standardized interpretation form
Sensitivity of SILVAMP-LAM versus the WHO symptom screening | 24-32 months
Area under the curve of SILVAMP-LAM versus the WHO symptom screening | 24-32 months
Specificity of SILVAMP-LAM versus the WHO symptom screening | 24-32 months
Sensitivity of Xpert Ultra performed on an oral/buccal swab versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Specificity of Xpert Ultra performed on an oral/buccal swab versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Area under the ROC curve of Xpert Ultra performed on an oral/buccal swab versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Sensitivity of Xpert Ultra performed on stool versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Specificity of Xpert Ultra performed on stool versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Area under the receiver operator curve of Xpert Ultra performed on stool versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Sensitivity of LF-LAM versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Specificity of LF-LAM versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Area under the receiver operator curve of LF-LAM versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Sensitivity of Xpert Ultra performed on a gelatin filter removed from a participant's mask versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Specificity of Xpert Ultra performed on a gelatin filter removed from a participant's mask versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Area under the receiver operator curve of Xpert Ultra performed on a gelatin filter removed from a participant's mask versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Sensitivity of point of care ultrasound versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Specificity of point of care ultrasound versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Area under the receiver operator curve of point of care ultrasound versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
Sensitivity of Xpert Host Response Cartridge on blood specimen versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
  The blood specimen is collected at the time of positive screening
Specificity of Xpert Host Response Cartridge on blood specimen versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
  The blood specimen is collected at the time of positive screening
Area under the receiver operator curve of Xpert Host Response Cartridge on blood specimen versus Xpert Ultra completed on sputum or gastric aspirate | 24-32 months
  The blood specimen is collected at the time of positive screening
Sensitivity of chest radiography for TB screening compared to the sensitivity of the WHO symptom screening using the McNemar test | 24-32 months
Sensitivity of SILVAMP-LAM for TB screening compared to the sensitivity of the WHO symptom screening using the McNemar test | 24-32 months

CONTACTS AND LOCATIONS:
Locations (5):
- Baylor College of Medicine Children's Foundation, Mbabane, Eswatini
- Baylor College of Medicine Children's Foundation, Maseru, Lesotho
- Baylor College of Medicine Children's Foundation, Lilongwe, Malawi
- Baylor College of Medicine Children's Foundation, Mbeya, Tanzania
- Baylor College of Medicine Children's Foundation, Kampala, Uganda